CLINICAL TRIAL: NCT03537586
Title: A Single Center Diagnostic, Cross-sectional Study of Coronary Microvascular Dysfunction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-00116
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Coronary Microvascular Disease; Ischemic Heart Disease; Myocardial Ischemia
MeSH Terms: conditions — Microvascular Angina; Myocardial Ischemia | interventions — bivalirudin; Adenosine; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-Obstructive CAD (Experimental): After diagnostic coronary angiography, invasive measures of coronary microvascular physiology will be obtained. Blood will be collected for platelet activity, inflammation and isolation of coronary endothelial cells.
  Interventions: Drug: Bivalirudin; Drug: Adenosine; Drug: Heparin; Device: Pressure-Temperature Sensor Guidewire; Device: Guiding Catheter

INTERVENTIONS:
Drug: Bivalirudin — After diagnostic catheterization, intravenous bivalirudin (Angiomax) will be administered as part of the research procedure, and a 6F-guiding catheter without side holes will be used to engage the ostium of the coronary artery.
  Other Names: Angiomax
Drug: Adenosine — An intravenous infusion of adenosine (140 μg/kg/min) will be administered via a large peripheral or central vein to induce steady-state maximal hyperemia.
  Other Names: Adenoscan
Drug: Heparin — Heparin may be used as an alternative to bivalirudin at the discretion of the interventional cardiologist.
Device: Pressure-Temperature Sensor Guidewire — Abbott's Pressure Wire X will be used to measure fractional flow reserve (FFR), cardiac magnetic resonance (CMR) and Index of Microcirculatory Resistance (IMR) in the Left Anterior Descending (LAD) Artery and major epicardial coronary vessels associated with myocardial ischemia.
  Other Names: Pressure Wire X
Device: Guiding Catheter — Medtronic's 6F Launcher Guide Catheter will be used to engage the left main coronary artery.
  Other Names: 6F Launcher Guide Catheter

SUMMARY:
Among patients with stable ischemic heart disease who are referred for coronary angiography, a substantial proportion have non-obstructive coronary artery disease (CAD). Ischemia based on symptoms or stress testing may be due to coronary microvascular dysfunction in up to 40% of these patients. However, the mechanisms and optimal treatment of coronary microvascular dysfunction are unknown. Aberrant platelet activity and inflammation have been hypothesized as mechanisms of microvascular dysfunction. Investigators plan to evaluate association between platelet activity, inflammation, and coronary microvascular dysfunction in stable women referred for coronary angiography, and to identify non-invasive correlates of coronary microvascular dysfunction in these patients.

DETAILED DESCRIPTION:
The objectives of this study are to

1. Investigate platelet activity and inflammation in patients with and without coronary microvascular disease who are referred for coronary angiography for the evaluation of stable ischemic heart disease and are found to have non-obstructuve epicardial CAD
2. To identify correlates of coronary microvascular dysfunction in non coronary microvascular beds that can be characterized in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Adult women age ≥18 years referred for coronary angiography
* Stable ischemic heart disease, defined by ischemic symptoms and/or myocardial ischemia by stress testing
* Administration of aspirin therapy prior to cardiac catheterization

Exclusion Criteria:

Pre-Cath Exclusion criteria:

* Active bleeding and/or bleeding diathesis
* Anemia (hemoglobin <9 mg/dl)
* Known thrombocytosis (platelet count >500,000)
* Know thrombocytopenia (platelet count <100,000)
* NSAIDs (e.g., ibuprofen, naproxen) within 3 days
* Platelet antagonists other than aspirin and thienopyridines, within 7 days
* Prior percutaneous coronary intervention or coronary artery bypass grafting
* Acute myocardial infarction within 3 months
* Severe valvular heart disease
* Cardiogenic shock or mechanical circulatory support
* New York Heart Association (NYHA) Functional Class III or IV heart failure
* Ejection Fraction <40%
* Hypertrophic obstructive cardiomyopathy or severe left ventricular hypertrophy
* Pregnancy
* Contraindication to intravenous infusion of adenosine during coronary angiography, due to known hypersensitivity to adenosine, known or suspected bronchoconstrictive or bronchospastic lung disease (severe asthma), second- or third-degree AV block (except in patients with a functioning artificial pacemaker), or sinus node disease, such as sick sinus syndrome or symptomatic bradycardia,

Angiographic Exclusion criteria:

* Obstructive CAD (≥50% luminal obstruction in ≥1 major epicardial coronary arteries by invasive coronary angiography)
* Unfavorable coronary artery anatomy for guidewire positioning (as determined by the angiographer or PI)

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Platelet Activity measured by the Index of Microcirculatory Resistance (IMR) | 12 Months
Measure of Inflammation measured by the Index of Microcirculatory Resistance (IMR) | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Smilowitz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Harkin KL, Loftspring E, Beaty W, Joa A, Serrano-Gomez C, Farid A, Hausvater A, Reynolds HR, Smilowitz NR. Visual Estimates of Coronary Slow Flow Are Not Associated With Invasive Wire-Based Diagnoses of Coronary Microvascular Dysfunction. Circ Cardiovasc Interv. 2024 Jun;17(6):e013902. doi: 10.1161/CIRCINTERVENTIONS.123.013902. Epub 2024 Apr 7. PMID 38583174